CLINICAL TRIAL: NCT04623814
Title: HEC113995-A Phase I,Double-Blind, Placebo-Controlled, Multiple Oral Dose, Safety, Tolerability, Pharmacokinetics and Food Effect Study in Healthy Chinese Subjects
Brief Title: the Safety, Tolerability, and Pharmacokinetics Study of HEC113995
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HEC113995-P-04/CRC-C2006
Record Dates: First submitted 2020-10-19; First posted 2020-11-10 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Food

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Food effect (Experimental): HEC113995 20mg will be administered fasted, with regular meal or with high-fat meal for once.
  Interventions: Other: Food
- Multiple Ascending Doses-HEC113995 10mg (Experimental): HEC113995 10mg will be administered fasted for 10 days
  Interventions: Drug: HEC113995
- Multiple Ascending Doses-HEC113995 20mg (Experimental): HEC113995 20mg will be administered with food for 10 days
  Interventions: Drug: HEC113995
- Multiple Ascending Doses-HEC113995 40mg (Experimental): HEC113995 40mg will be administered with food for 10 days
  Interventions: Drug: HEC113995
- Multiple Ascending Doses-placebo (Placebo Comparator): Placebo arms will be administered fasted or with food for 10 days
  Interventions: Drug: placebo

INTERVENTIONS:
Other: Food — HEC113995 20mg will be taken orally fasted or with food
  Arms: Food effect
Drug: HEC113995 — HEC113995 will be taken orally fasted (HEC113995 10mg）or with food (HEC113995 20mg and 40mg） for 10 days
  Arms: Multiple Ascending Doses-HEC113995 10mg; Multiple Ascending Doses-HEC113995 20mg; Multiple Ascending Doses-HEC113995 40mg
Drug: placebo — The placebo will be administered fasted or with food for 10 days.
  Arms: Multiple Ascending Doses-placebo

SUMMARY:
Multiple Dose Safety, Tolerability, PK and Food Effect Study of HEC113995 PA•H2O in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects who are willing and are able to provide a written informed consent to participate in the study.
* 2. Without Plan for pregnancy or pregnant within 3 months after enrollment throughout the trial.
* 3. Subjects aged between 18 and 45 (both inclusive) years old.
* 4. Healthy volunteers has a body weight ≥50 kg (for male) or ≥ 45kg (for female) and body mass index ≥18 and ≤28 kg/m2 at screening.
* 5. Subjects, who are healthy, as having no clinically significant abnormalities in vital signs, physical examination, clinical laboratory test results, Chest X-ray and 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* 1. Subjects with a positive serology for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies and/or TP antibodies at screening.
* 2. Subjects with history of digestive system,urinary system, liver,central nervous system, blood system, endocrine system,respiratory system,immune system,cardiovascular system,and/or malignant tumor or others medical conditions (such as history of mental illness, etc.) that are not suitable for clinical trial participation;Subjects with history of epilepsy, bipolar disorder/mania, high intraocular pressure, or acute angular-closure glaucoma.
* 3. Known allergic reactions or hypersensitivity to any excipient of the drug formulation(s) ,or anaphylaxis physique.
* 4. Use of any prescription or non-prescription medications within 14 days prior to initial dosing,or Use of any medications known to inhibit or induce cytochrome P enzyme drug metabolism within 28 days prior to initial dosing.
* 5. Consume foods or beverages containing caffeine, xanthine, alcohol, and grapefruit within 48 hours prior to initial dosing.
* 6. Positive results from urine drug screen test.
* 7. History of alcoholism or drink regularly within 3 months prior to the study(defined as Alcohol consumption of > 21 units/week), or positive results from alcohol breath test.
* 8. Regular smoking of more than 10 cigarettes per day within 3 months before administration of study drug.
* 9. Donate blood or lose blood 400 mL or more within 1 month prior to initial dosing.
* 10. Subjects who plan to receive or have had organ transplants.
* 11. Females who are lactating/breastfeeding, or positive result from pregnancy test for women of child-bearing potential.
* 12. Subjects who participated in another clinical trial within 3 months prior to initial dosing.
* 13. Any other condition with in the opinion of the investigator would render the patient unsuitable for inclusion in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Adverse event | up to 34 days
  To assess the safety and tolerability of therapy

SECONDARY OUTCOMES:
Area under the concentration versus time curve (AUC) from time zero to infinity(AUC0-∞ ) | up to 120 hours
Maximum Plasma Concentration （ Cmax） | up to 120 hours
Time to peak（tmax） | up to 120 hours
Apparent terminal elimination half-life（t½） | up to 120 hours
Apparent volume of distribution（Vz/F） | up to 120 hours
The Mean Residence Time（ MRT） | up to 120 hours
The Apparent Clearance （CL/F） | up to 120 hours
The Accumulation Ratio（R） | up to 120 hours
Food Effect on the Cmax | up to 120 hours
Food Effect on the AUC | up to 120 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No